CLINICAL TRIAL: NCT05669690
Title: The Effect of Storage Conditions on Microbiota Composition of Breast Milk
Brief Title: Storage Conditions and Breast Milk Microbiota Composition
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Beril Yasa, Assistant Professor, Istanbul University
Other Study IDs: 39040
Record Dates: First submitted 2022-12-20; First posted 2023-01-03 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Breast Milk Collection; Microbial Colonization
Keywords: breast milk; storage conditions; microbiota
MeSH Terms: conditions — Breast Milk Expression; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Breast milk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Fresh breast milk: Fresh breast milk obtained from volunteer mothers will be divided into four parts. Fresh breast milk will be studied for microbiota composition immediately within 3 hours.
- Breast milk stored at +4'C for 3 days: One part of previously obtained fresh breast milk will be stored at +4'C at refrigerator for 3 days long, then microbiota composition will be studied.
- Breast milk stored at -20'C for 3 months: Last part of the same breast milk specimen will be freezed at -20'C for 3 months and microbiota composition of the 3 months frozen milk will be studied.

SUMMARY:
Breast milk is the mainstay of newborn nutrition, providing all the nutrients and vitamins necessary for optimal growth of newborn infants. Beside its nutritional properties, breast milk also contains bioactive factors such as soluble immune factors, antimicrobial proteins, functional fatty acids, hormones, oligosaccharides, stem cells and microbiota. Although fresh breast milk is the optimal source of nutrition for newborn infants, breast milk must be expressed and stored in some conditions.

Breast milk was thought to be sterile for many years. This idea has changed with the isolation of live bacteria in the breast milk of healthy mothers in the recent past. Thus, it has been shown that breast milk is not actually a sterile body fluid, but has a microbiota of its own. This study aimed to examine the effect of storage conditions of breast milk at different temperatures on the microbial composition of the breast milk.

The prospective experimental study will be conducted under the supervision of Istanbul University, Istanbul Medical Faculty, Department of Pediatrics, Neonatology Department. Informed consent of mothers will be taken. Thirty mililiter (30 mL) breast milk that was obtained from volunteer mothers will be divided into 3 samples, each 10 mL of breast milk will be stored at different temperatures. Ten mililiter will be studied for microbial composition with 16S rRNA amplicon sequencing and bioinformatics analysis immediately, 10 mL will be stored at +4'C for 3 days and will be studied at the end of 3rd day, other 10 mL will be stored at -20'C for 3 months and will be studied at the end of 3rd months. 16S rRNA amplicon sequencing and bioinformatic analysis studies will be performed at Istanbul Medical Faculty Clinical Nutrition and Microbiota Research Laboratory.

This present study is planned to be carried out for 24 months between January 2023 and December 2024

DETAILED DESCRIPTION:
Fresh breast milk is the mainstay of newborn nutrition and provides all the nutrients and vitamins needed for optimal growth of newborn babies. In addition to the nutritional properties of breast milk, there are some bioactive factors such as soluble immune factors, antimicrobial proteins, functional fatty acids, hormones, oligosaccharides, stem cells and microbiota in breast milk. Breastfeeding also strengthens the bond between mother and baby in postpartum period and provides nutrition to the newborn infant. Breast milk improves microbial colonization, improves immune system maturation and supports the metabolic activities of the newborn infant.

Although fresh breast milk is the optimal food source for newborn babies, in some cases, breast milk must be expressed and stored.It is reported that breast milk can be stored in the refrigerator for 3 days without being frozen at +4 degrees Celsius, and can be stored as frozen for 3 months if it is frozen within the first 24 hours after milking. The North American Breast Milk Banking Association, on the other hand, reports that the storage period can be extended up to 12 months at temperatures below -20 degrees Celsius.

While breast milk was thought to be a sterile fluid, this idea has changed with the isolation of live bacteria in the milk of healthy mothers in the recent past. The presence of many bacteria such as Lactobacillus, Lactococcus, Bifidobacterium, Streptococcus, Enterococcus and Staphylococcus has been demonstrated by traditional culture methods of breast milk. The new generation sequencing technologies obtained higher microbial diversity of breast milk and detected mouth-dwelling bacteria such as Veillonella and Prevotella, skin bacteria such as Propionobacterium and gram-negative bacteria such as Pseudomonas, Ralstonia, Klebsiella. Thus, it has been shown that breast milk is not actually a sterile body fluid, but has a microbiota of its own.

There are few studies evaluating the effect of breast milk storage conditions on microbiota. In a study, it was shown that the number of bacterial colonies in breast milk decreased as the freezing period increased. It has been shown that 98-100% of bacteria in frozen breast milk are lost after 12 weeks of storage.

Although studies evaluating fresh breast milk microbiota have been reported in the literature, there are few studies evaluating the effect of milk storage conditions on microbial diversity. In existing studies, microbial growth was ensured by culture method and diversity was defined by traditional microbiological methods. No study was found that evaluated the microbial composition of breast milk with next-generation sequencing based on the 16S rRNA amplicon sequencing strategy.

This study aimed to evaluate how the generally recommended breast milk storage conditions and duration of storage affect the microbiota composition of breast milk. This study will provide new data and new recommendations about storage of breast milk.

ELIGIBILITY:
Inclusion Criteria:

* Women who had vaginal delivery
* Women who gave delivery at gestational age above 37 weeks
* Women who have a child older than 1 weeks of age
* Mothers with a body mass index between 18.5-25
* Women who gave consent

Exclusion Criteria:

* Women who had cesarean delivery
* Women who gave premature delivery (<37 weeks of gestation)
* Women who gave birth within prior 7 days
* Women with premature rupture of membranes
* Women with chorioamnionitis
* Women who had antibiotherapy within last 1 week
* Presence of mastitis
* Presence of maternal co-morbid diseases such as; pregestational diabetes, pregestational hypertension, connective tissue diseases, inflammatory bowel syndrome, solid organ transplantation
* Presence of evidenced congenital infections
* Women who didn't give consent

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy young mothers who had vaginal delivery at least one week ago will be included
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2024-12-14 (Estimated)

PRIMARY OUTCOMES:
Changes in microbiota composition of breast milk after storage | 24 months
  To evaluate the effects of different storage conditions on microbiota composition of breast milk

CONTACTS AND LOCATIONS:
Overall Officials: Emine Asuman Coban, Professor, Principal Investigator — Istanbul University; Elmas Zeynep Ince, Professor, Principal Investigator — Istanbul University; Bülent Saka, Professor, Principal Investigator — Istanbul University; Leyla Bilgin, Professor, Principal Investigator — Istanbul University; Dilek Sever Kaya, Dr Biologist, Principal Investigator — Istanbul University; Aslı Berru Arslan, Med Student, Principal Investigator — Istanbul University; Beril Yasa, Ass. Prof., Study Director — Istanbul University
Locations (1):
- Istanbul University Istanbul Medical Faculty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
It is planned to share individual participant data in terms of changes in microbiota composition of breast milk with different storage conditions. Special data about identity of participants will be kept blinded.
Supporting Information: CSR
Time Frame: Data about Clinical Study Report will become available after all samples are obtained, analyzed and study completed. The data will be available for 12 months period.
Access Criteria: The IPD will be uploaded to the registration system, any investigator will be able to access IPD

REFERENCES:
- [Background] Selma-Royo M, Calvo Lerma J, Cortes-Macias E, Collado MC. Human milk microbiome: From actual knowledge to future perspective. Semin Perinatol. 2021 Oct;45(6):151450. doi: 10.1016/j.semperi.2021.151450. Epub 2021 Jun 16. PMID 34274151
- [Background] Pandya SP, Doshi H, Codipilly CN, Fireizen Y, Potak D, Schanler RJ. Bacterial stability with freezer storage of human milk. J Perinat Med. 2020 Sep 14;49(2):225-228. doi: 10.1515/jpm-2020-0131. Print 2021 Feb 23. PMID 32915767
- [Result] Fernandez L, Ruiz L, Jara J, Orgaz B, Rodriguez JM. Strategies for the Preservation, Restoration and Modulation of the Human Milk Microbiota. Implications for Human Milk Banks and Neonatal Intensive Care Units. Front Microbiol. 2018 Nov 9;9:2676. doi: 10.3389/fmicb.2018.02676. eCollection 2018. PMID 30473683